CLINICAL TRIAL: NCT00801684
Title: Efficacy, Safety, Tolerability, and Pharmacokinetics of Trospium Inhalation Powder (TrIP) Administered to Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: ALK27-001: A Study of Trospium Inhalation Powder (TrIP)Administered to Subjects With COPD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Bernard L. Silverman, MD / VP, Clinical Development, Alkermes, Inc.
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALK27-001
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Results first posted 2011-05-10 (Estimated); Last update posted 2011-08-19 (Estimated); Status verified 2011-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; pulmonary; inhalation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Placebo (Placebo Comparator): Represents Dose A in the Dosing Sequence assignments.
  Interventions: Drug: Placebo
- TrIP-2D (100mcg) (Experimental): Represents Dose B
  Interventions: Drug: TrIP-2D
- TrIP-2SS (100mcg) (Experimental): Represents Dose C
  Interventions: Drug: TrIP-2SS
- TrIP-2D (400mcg) (Experimental): Represents Dose D
  Interventions: Drug: TrIP-2D
- TrIP-2SS (100mcg) + Foradil (12mcg) (Experimental): Represents Dose E. All subjects received Dose E as their final (5th) dose, after completing their initial 4 single doses according to their sequence assignment.
  Interventions: Drug: TrIP-2SS + Foradil

INTERVENTIONS:
Drug: Placebo — Supplied as an empty size-2 capsule and administered as a single dose via C2S inhaler.
  Arms: Placebo
Drug: TrIP-2D — Trospium inhalation powder containing 100 mcg TrCl (trospium chloride), supplied as dry powder in size-2 capsules and administered as a single dose via C2S inhaler.
  Arms: TrIP-2D (100mcg)
Drug: TrIP-2SS — Trospium inhalation powder containing 100 mcg TrCl (trospium chloride), supplied as dry powder in size-2 capsules and administered as a single dose via C2S inhaler.
  Arms: TrIP-2SS (100mcg)
Drug: TrIP-2D — Trospium inhalation powder containing 400 mcg TrCl (trospium chloride), supplied as dry powder in size-2 capsules and administered as a single dose via C2S inhaler.
  Arms: TrIP-2D (400mcg)
Drug: TrIP-2SS + Foradil — Trospium inhalation powder containing 100 mcg TrCl (trospium chloride), plus foradil (12 mcg formoterol fumarate) supplied as dry powder in size-2 capsules and administered as a single dose via C2S inhaler.
  Arms: TrIP-2SS (100mcg) + Foradil (12mcg)

SUMMARY:
The purpose of this study was to evaluate the efficacy, safety, and tolerability of single doses of trospium inhalation powder (TrIP) administered to subjects with chronic obstructive pulmonary disease (COPD).

DETAILED DESCRIPTION:
This was a single-center, randomized, double-blind, cross-over, placebo-controlled study. Following screening, each eligible subject was randomized to a dosing sequence. Study subjects received a total of 5 single doses, each separated by a 3- to 14-day washout period. Doses A, B, C, and D were administered in a double-blind fashion, in sequences generated by a 4-period Latin square design. The 4 dosing sequences were: ABCD, BDAC, CADB, and DCBA. Dose E was administered in an open-label fashion as the final dose in each dosing sequence for all subjects.

Subjects reported to the clinic the evening prior to each dose. Protocol assessments were carried out until 24 hours postdose. Pulmonary function testing (via spirometry) was captured at specified timepoints at baseline as well as before and after dosing. Other efficacy and safety outcomes were assessed according to protocol. Blood sampling was performed for assessment of trospium concentrations at specified timepoints.

ELIGIBILITY:
Inclusion Criteria:

* Male or female COPD subjects between the ages of 40 and 80 years
* Body mass index between 18 and 35
* Medically healthy (other than COPD)
* FEV1/FVC less than or equal to 0.70
* Current non-smoker or able to abstain from smoking for at least 8 hours postdose
* Within the previous 6 months, demonstrated improvement in FEV1 (greater than or equal to 10%) 1 hour following administration of ipratropium bromide inhalation (4 puffs)
* Females of childbearing potential must agree to use an acceptable method of contraception for the duration of the study

Exclusion Criteria:

* Asthma in the last 10 years
* Allergic rhinitis, atopy, cystic fibrosis, bronchiectasis, or tuberculosis
* Bladder neck obstruction, including urinary retention or known symptomatic prostatic hypertrophy not controlled with medication
* Narrow angle glaucoma
* Tachyarrhythmia
* Alcohol dependence or illicit drug abuse within the past year
* Using long-term oxygen therapy
* Female subjects who are pregnant or breastfeeding
* Participating in another clinical trial

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bernard L. Silverman, MD, Study Director — Alkermes, Inc.
Locations (1):
- Spartanburg Medical Research, Spartanburg, South Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Overall Study: Following screening, each subject was randomized to a sequence of 5 dosing periods (Doses A, B, C, D, and E). Each period was separated by a 3- to 14-day washout interval. Doses A, B, C, and D were administered in a double-blind fashion. Dose E was administered in an open-label fashion.
  The dosing formulations were as follows:
  Dose A = placebo Dose B = TrIP-2D (100 μg TrCl formulated in leucine and DPPC) Dose C = TrIP-2SS (100 μg TrCl formulated in leucine and sodium saccharin) Dose D = TrIP-2D (400 μg TrCl) Dose E = TrIP-2SS (100 μg TrCl) + Foradil (12 μg formoterol fumarate)
Period: Overall Study
Arm/Group | Overall Study
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Overall Study
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 9
Age Continuous [Mean (Standard Deviation); unit: years] | 63.0 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Spirometry Parameter: Peak Forced Expiratory Volume in 1 Second(FEV1)in Liters (L)
Description: Following screening, each subject was randomized to a sequence of 5 dosing periods (Doses A, B, C, D, and E). Each period was separated by a 3- to 14-day washout interval.
  The dosing formulations were as follows:
  Dose A = placebo Dose B = TrIP-2D (100 μg TrCl formulated in leucine and DPPC) Dose C = TrIP-2SS (100 μg TrCl formulated in leucine and sodium saccharin) Dose D = TrIP-2D (400 μg TrCl) Dose E = TrIP-2SS (100 μg TrCl) + Foradil (12 μg formoterol fumarate) FEV1 (L)was measured at 15 and 30 minutes, 1, 2, 3, 4, 6, 8, 12 and 24 hours postdose.
Time Frame: 15 minutes to 24 hours post-treatment
Measure: Mean (Standard Deviation); unit: Liters
Groups:
- TrIP-2SS (100mcg): Subjects were administered TrIP (100mcg) over 5 dosing periods, each separated by a 3- to 14 day washout period. Subjects reported to the clinic the evening prior to each dose, and assessments were carried out through 24 hours postdose. A 3- to 14-day washout period was maintained between doses. Trospium inhalation powder containing 2% TrCl (100 mcg) formulated in leucine and sodium saccharin, supplied as dry powder in size-2 capsules, was administered via a dry powder inhaler.
- TrIP-2SS (100mcg) + Foradil (12mcg): Subjects were administered TrIP (100mcg)plus Foradil (12mcg)over 5 dosing periods, each separated by a 3- to 14 day washout period. Subjects reported to the clinic the evening prior to each dose, and assessments were carried out through 24 hours postdose. A 3- to 14-day washout period was maintained between doses. Foradil (12mcg)and Trospium inhalation powder containing 2% TrCl (100 mcg) formulated in leucine and sodium saccharin, supplied as dry powder in size-2 capsules, was administered via a dry powder inhaler.
- TrIP-2D (100mcg): Subjects were administered TrIP-2D (100mcg) over 5 dosing periods, each separated by a 3- to 14 day washout period. Subjects reported to the clinic the evening prior to each dose, and assessments were carried out through 24 hours postdose. A 3- to 14-day washout period was maintained between doses. Trospium inhalation powder containing 2% TrCl (100 mcg) formulated in leucine and DPPC; supplied as dry powder in size-2 capsules and administered via dry powder inhaler. One capsule (100 mcg TrCl) or 4 capsules (400 mcg TrCl) were used. A separate inhaler was provided for each capsule.
- TrIP-2D (400mcg): Subjects were administered TrIP-2D (400mcg)over 5 dosing periods, each separated by a 3- to 14 day washout period. Subjects reported to the clinic the evening prior to each dose, and assessments were carried out through 24 hours postdose. A 3- to 14-day washout period was maintained between doses. Trospium inhalation powder containing 2% TrCl (100 μg) formulated in leucine and DPPC; supplied as dry powder in size-2 capsules and administered via dry powder inhaler. One capsule (100 μg TrCl) or 4 capsules (400 μg TrCl) were used. A separate inhaler was provided for each capsule.
- Placebo: Subjects were administered placebo over 5 dosing periods, each separated by a 3- to 14 day washout period. Subjects reported to the clinic the evening prior to each dose, and assessments were carried out through 24 hours postdose. A 3- to 14-day washout period was maintained between doses. Placebo was supplied as empty Size-2 capsules and administered via a dry powder inhaler.
Arm/Group | TrIP-2SS (100mcg) | TrIP-2SS (100mcg) + Foradil (12mcg) | TrIP-2D (100mcg) | TrIP-2D (400mcg) | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Liters | 1.707 (0.528) | 1.696 (0.521) | 1.672 (0.528) | 1.676 (0.516) | 1.508 (0.545)
Statistical Analysis 1: Comparison: TrIP-2SS (100mcg) vs TrIP-2SS (100mcg) + Foradil (12mcg) vs TrIP-2D (100mcg) vs TrIP-2D (400mcg) vs Placebo; The difference between the active treatment was compared to placebo. For a null hypothesis, the difference would equal 0 (zero); Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: FEV1 Response to Treatment
Description: Response was defined as the number of subjects reporting a post-treatment FEV1 of ≥12% (or 200 mL) above baseline.
Time Frame: Up to 24 hours post-treatment
Population: All 24 randomized subjects were included in the analysis.
Measure: Number; unit: Participants
Arm/Group | TrIP-2SS (100mcg) | TrIP-2SS (100mcg) + Foradil (12mcg) | TrIP-2D (100mcg) | TrIP-2D (400mcg) | Placebo
Number analyzed (Participants) | 24 | 24 | 24 | 24 | 24
Participants | 23 | 22 | 22 | 21 | 14

3. Secondary Outcome: Time to Maximum Plasma Concentration (Tmax) of Trospium After Single Administrations of TrIP
Description: Tmax is reported as median (range) of hours to reach maximum trospium concentration in plasma.
Time Frame: up to 24 hours post-treatment
Population: The PK population consisted of all subjects who received active study medication and had sufficient concentration data to facilitate calculation of the PK parameters or descriptive statistics of concentrations of trospium.
Measure: Median (Full Range); unit: Hours
Groups:
- TrIP-2D (400mcg): Subjects were administered TrIP-2D (100mcg) over 5 dosing periods, each separated by a 3- to 14 day washout period. Subjects reported to the clinic the evening prior to each dose, and assessments were carried out through 24 hours postdose. A 3- to 14-day washout period was maintained between doses. Trospium inhalation powder containing 2% TrCl (100 mcg) formulated in leucine and DPPC; supplied as dry powder in size-2 capsules and administered via dry powder inhaler. One capsule (100 mcg TrCl) or 4 capsules (400 mcg TrCl) were used. A separate inhaler was provided for each capsule.
Arm/Group | TrIP-2D (100mcg) | TrIP-2SS (100mcg) | TrIP-2D (400mcg) | TrIP-2SS (100mcg) + Foradil (12mcg)
Number analyzed (Participants) | 12 | 12 | 12 | 24
Hours | 0.08 [0.03 to 0.08] | 0.08 [0.02 to 0.48] | 0.08 [0.03 to 0.08] | 0.08 [0.02 to 0.52]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored continuously from the time the subject signed the consent form until the end of the last dosing period.
Arm/Group | Overall Study | TrIP-2D (100mcg) | TrIP-2SS (100mcg) | TrIP-2D (400mcg) | TrIP-2SS (100mcg) + Foradil (12mcg) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 6/24 | 1/24 | 2/24 | 4/24 | 1/24 | 1/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Overall Study (N=24) | TrIP-2D (100mcg) (N=24) | TrIP-2SS (100mcg) (N=24) | TrIP-2D (400mcg) (N=24) | TrIP-2SS (100mcg) + Foradil (12mcg) (N=24) | Placebo (N=24)
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 1 | 0 | 0
Viral infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 1 | 1 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No individual Investigator may publish results without written agreement from Alkermes. Should an Investigator wish to publish or present the data at a meeting, a copy of the manuscript or abstract must be provided to the Sponsor at least 30 days prior to the submission for review and approval. Any revisions will be negotiated in good faith by the Investigator and Sponsor.